CLINICAL TRIAL: NCT01086865
Title: Clinical Study Phase III, Randomized, Double-blind, Prospective and Comparative to Evaluate the Efficacy and Tolerability of Using APETIVITON BC Compared to Petivit BC in Appetite Stimulate.
Acronym: Apetiviton BC
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cifarma Cientifica Farmaceutica Ltda (Industry)
Responsible Party: Sônia Silveira Braga, Cifarma Cientifica Farmaceutica Ltda
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: E02-CIF-APE-02-08
Record Dates: First submitted 2010-03-12; First posted 2010-03-15 (Estimated); Last update posted 2010-05-19 (Estimated); Status verified 2009-03

CONDITIONS: Inappetence
Keywords: inappetence; apetiviton BC
MeSH Terms: conditions — Anorexia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Petivit BC (Active Comparator)
  Interventions: Drug: Apetiviton BC
- Apetiviton BC (Experimental)
  Interventions: Drug: Apetiviton BC

INTERVENTIONS:
Drug: Apetiviton BC — Administer the recommended dosage preferably one hour before the main meal:
  Children (2 to 6 years): 2.5 mL 3 x daily. Adults (18 to 50 years): 5 mL 3 x daily. Elderly (60 to 80 years): 5 ml 3 x daily.
  Other Names: Petivit Bc

SUMMARY:
Clinical study phase III, randomized, double-blind, prospective, comparative non-inferiority to evaluate the efficacy and tolerability of using APETIVITON BC compared to Petivit BC in appetite stimulate in children, adults and elderly.

DETAILED DESCRIPTION:
Clinical trial phase III, randomized, double-blind, prospective, comparative non-inferiority to evaluate the efficacy and tolerability of using APETIVITON BC compared to Petivit BC stimulation of appetite in children, adults and elderly. A total of 150 patients, distributed as follows:

25 patients treated children Apetiviton BC,25 patients treated children Petivit BC, (2-6 years).

25 adult patients treated with Apetiviton BC,25 adult patients treated with Petivit BC, (18-50 years.

25 elderly patients treated with Apetiviton BC,25 elderly patients treated with Petivit BC. (60-80 years.

ELIGIBILITY:
Inclusion Criteria:

For both groups:

* Patients who have inappetence;
* Patients able to understand and maintain adherence to protocol;
* Wash-out 20 days after ingestion of prior similar drug;
* Patients able to understand the correct use of medication;
* Patients who consent to participate in the study by signing the inform consent;

Children:

* Patients of any ethnic group male and female, aged between 2 and 6 years;

Adults:

* Patients of any ethnic group male and female, aged between 18 and 50 years;
* Female patients in childbearing age, sexually active, make pregnancy test result should be negative and, furthermore, should be using contraceptive methods such as contraception, condom, IUD and diaphragm.

Elderly:

* Patients of any ethnic group male and female, aged between 60 and 80 years.
* Female patients in childbearing age, sexually active, make pregnancy test result should be negative and, furthermore, should be using contraceptive methods such as contraception, condom, IUD and diaphragm.

Exclusion Criteria:

For both groups:

* Patients with glaucoma open or closure angle;
* Patients with predisposition to urinary retention;
* Patients with stenous peptic ulcer or pylorus-duodenal obstruction;
* Debilitated patients or in acute attack of asthma;
* Alcoholic;
* Patients who have loss of appetite caused by any serious disease;
* Patients who make use of any drugs central nervous system depressants;
* Patients who make use of medicines monoaminooxidase inhibitors, tricyclic antidepressants, phenothiazines, probenecid, levodopa, phenytoin, phenobarbital, chloramphenicol, cyclophosphamide, cyclosporine, chlorambucil, corticotropin, mercaptopurine, isoniazid, penicillin, estrogens, contraceptives, haloperidol, ipatrópico, barbiturates, primidone, salicylates;
* Patients with known hypersensitivity to any components of the formula;
* Patient who is participating in another clinical study;
* No able to adhere to protocol;
* Patients who are pregnant or breastfeeding;
* Any condition that in the opinion of the investigator can impossible to include the patient's adherence to the protocol.

Ages: 2 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2010-08; Primary Completion 2010-11 (Estimated); Study Completion 2011-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effectiveness of apetiviton BC compared to Petivit BC in appetite stimulation in children, adults and seniors. | 30 days

SECONDARY OUTCOMES:
Evaluate the tolerability of apetiviton BC compared to Petivit BC the stimulation of appetite in children, adults and seniors | 30 days